CLINICAL TRIAL: NCT06100770
Title: Aveir AR Coverage With Evidence Development (CED) Study
Acronym: ARRIVE
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-CL1021378
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Pacemaker; Arrhythmia; Bradycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Aveir AR Leadless Pacemaker: This study will utilize real-world data from patients implanted with the Aveir AR Leadless Pacemaker. No device intervention is required in this study.
  Interventions: Device: Aveir AR Leadless Pacemaker
- Single-Chamber Atrial Transvenous Pacemaker: This study will utilize real-world data from patients implanted with a single-chamber atrial transvenous pacemaker as a comparator to the Aveir AR LP study arm. No device intervention is required in this study.
  Interventions: Device: Single-chamber atrial transvenous pacemaker

INTERVENTIONS:
Device: Aveir AR Leadless Pacemaker — This study will utilize real-world data from patients implanted with the Aveir AR Leadless Pacemaker. No device intervention is required in this study.
  Groups: Aveir AR Leadless Pacemaker
Device: Single-chamber atrial transvenous pacemaker — This study will utilize real-world data from patients implanted with a single-chamber atrial transvenous pacemaker as a comparator to the Aveir AR LP study arm. No device intervention is required in this study
  Groups: Single-Chamber Atrial Transvenous Pacemaker

SUMMARY:
The purpose of this coverage with evidence development (CED) study is to evaluate complications and long-term health outcomes of the single-chamber Aveir Atrial Leadless Pacemaker device (aka Aveir™ AR LP system).

DETAILED DESCRIPTION:
This CED study utilizes a real-world evidence (RWE) method merging multiple real-world datasets from Abbott and the Center for Medicare Services to assess Aveir AR LP health outcomes among Medicare beneficiaries.

The study will enroll all Medicare patients with continuous claims data implanted with the Aveir AR LP or a single-chamber atrial transvenous pacemaker system from any manufacturer.

Due to the RWE data collection methods used in this study, a central institutional review board (IRB) approved informed consent waiver has been granted. Due to this waiver and the sponsor's use of the central IRB, individual hospitals are not required to consent patients or complete local IRB submissions for this RWE study.

ELIGIBILITY:
Inclusion Criteria:

1. Medicare beneficiaries implanted with an Aveir AR leadless pacemaker on or after the study start date (i.e., the date of Aveir AR market approval) will be included in the study.

   OR
2. Medicare beneficiaries implanted with a full system (e.g. lead and generator) single chamber atrial transvenous pacemaker on or after the study start date

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include all Medicare patients with continuous claims data implanted with an Aveir DR leadless pacemaker or a full-system dual-chamber transvenous pacemaker (from any manufacturer) in any US location.
Sampling Method: Non-Probability Sample
Enrollment: 586 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Acute device-related complication rate | 30 days
  Assess the acute (30-day) complication rate of the Aveir AR LP, compared to single chamber atrial transvenous pacemakers. An acute complication is defined as a peri-procedural, device-related adverse event occurring within 30 days post-implant.
Two-year survival rate | 2 years
  Assess (2-year) survival rate of subjects implanted with an Aveir AR LP, compared to single chamber atrial transvenous pacemakers.

SECONDARY OUTCOMES:
Chronic complication rate | 6 months
  • To assess the chronic (6-month) complication rate of the Aveir AR LP, compared to single chamber atrial transvenous pacemakers. A chronic complication is defined as a post-procedural, device-related adverse event that requires invasive intervention to resolve, occurring more than 30 days through six months post implant.
Device related re-intervention rate | 2 years
  • To assess (2-year) device-related re-intervention rates of the Aveir AR LP, compared to single chamber atrial transvenous pacemakers.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (1):
- Abbott, Sylmar, California, United States